CLINICAL TRIAL: NCT04212403
Title: A Prospective Study About the Safety of Omitting Antibiotic Prophylaxis in Transurethral Prostate Resection (TURP) and Transurethral Bladder Tumour Resection (TURB): the prophylaxis001-trial
Brief Title: Antibiotic Prophylaxis in Transurethral Prostate Resection (TURP) and Transurethral Bladder Tumour Resection (TURB)
Acronym: Prophylaxis001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JessaH_B243201733480
Record Dates: First submitted 2019-08-06; First posted 2019-12-27 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Urosepsis; Bladder Cancer; Prostate Hyperplasia; Antibiotic Resistant Strain; Antibiotic Resistant Infection; Antibiotic-associated Diarrhea; Antibiotic Toxicity
Keywords: TURP; TURB
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Hyperplasia | interventions — Levofloxacin

STUDY DESIGN:
Intervention Model Description: Randomized, controlled trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): The control groups receives antimicrobial prophylaxis (AMP) as recommended by the guidelines.
  Interventions: Drug: Levofloxacin
- Treatment group (No Intervention): The treatment group receives no AMP.

INTERVENTIONS:
Drug: Levofloxacin — The control group receives AMP.
  Arms: Control

SUMMARY:
To investigate the use of antibiotic prophylaxis in patients undergoing TURP and TURB. The investigators set up a prospective, randomized controlled trial in which (after exclusion of risk factors) patients will be randomized in receiving levofloxacin (Tavanic) orally or no antibiotics. The exclusion criteria for TURP are a pre-operative transurethral catheter or > 100 urinary white blood cells in the pre-operative urine sample. The exclusion criteria for TURB are a pre-op catheter or clinical signs of infection.

DETAILED DESCRIPTION:
Main objective:

To investigate the safety of omitting antibiotic prophylaxis in TURP (transurethral resection of the prostate) and TURB (transurethral bladder tumour resection) in patients without a pre-operative catheter or > 100 WBC in the pre-operative urinary sample (TURP) or clinical signs of urinary infection (TURB).

Secondary objective:

To investigate post-operative bacteriuria after TURB and TURP in our population.

Principal inclusion criterium:

Patients undergoing TURP or TURB.

Primary exclusion criterium:

TURP: pre-operative catheter or > 100 white blood cells in the pre- operative urinary sample.

TURB: pre-operative catheter or clinical signs of infection (fever, nyctalgia).

Primary endpoint:

Post-operative infection.

Secondary endpoint:

Post-operative bacteriuria.

ELIGIBILITY:
Inclusion Criteria:

* TURP or TURB.

Exclusion Criteria:

* TURP: pre-operative catheter/DJ/nephrostomy or > 100 white blood cells in the pre- operative urinary sample.

TURB: pre-operative catheter/DJ/nephrostomy or clinical signs of infection (fever, myctalgia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1350 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
% of patients with a post-operative infection. | From immediately post-op until at the control consultation 4 weeks after surgery.
  Urosepsis, fever (t°> 38.5) or epididymitis.

SECONDARY OUTCOMES:
Incidence of post-operative bacteriuria. | From immediately post-op until at the control consultation 4 weeks after surgery.
  > 100.000 bacteria/mL urine

CONTACTS AND LOCATIONS:
Overall Officials: Koenraad van Renterghem, PhD, Principal Investigator — UHasselt
Locations (1):
- Jessa Ziekenhuis, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided